CLINICAL TRIAL: NCT06873061
Title: Principal Investigator, Doktor Researcher Assistant, Department of Psychiatric Nursing
Brief Title: "The Impact of Digitalization Education Provided to Nursing Students on Their Attitudes Towards Telemedicine"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Kubra Gulırmak, Dr. Researcher, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024-384
Record Dates: First submitted 2025-03-04; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Telenursing; Telemedicine
Keywords: telemedicine; telenursing; nursing student
MeSH Terms: interventions — Telenursing

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial (RCT) is a research design in which participants are randomly assigned to either an experimental group or a control group. The experimental group receives a specific intervention or treatment, while the control group receives no intervention or the standard treatment. In this way, the effect of the intervention is assessed. Pre- and post-intervention data are collected, and the differences between the groups are evaluated using statistical analysis. RCT is a reliable method for objectively measuring the effects of an intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): During the study, no intervention was applied to the students in the control group, except for the pre-test and post-test measurements.
- experimental group (Experimental): The students in the experimental group underwent pre-test and post-test assessments and received telemedicine training for 5 weeks.
  Interventions: Other: telenursing

INTERVENTIONS:
Other: telenursing — This study aims to examine the impact of telemedicine training on nursing students. The training content is designed specifically for nursing students and includes various techniques such as simulations.
  Arms: experimental group

SUMMARY:
This research was conducted as a pre-test post-test design in a randomized controlled study. Participants were given a 5-week telemedicine education related to nursing care, and the changes in students' attitudes toward telemedicine were examined. Digitalization has brought about significant changes in healthcare, and telemedicine applications have enabled nurses to transform patient care. Improving nursing students' knowledge and attitudes toward telehealth is crucial for enhancing the effective use of digital health tools. In this context, the "The Role of Digitalization in Nursing: An Innovative Transformation in Care" training program was designed to assess nursing students' attitudes toward telemedicine applications. The study aims to analyze the impact of the training program by comparing experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older,
* Currently enrolled as an active student in the Nursing Department,
* A third-year student in the Nursing Department,
* Agreement to participate in the study.

Exclusion Criteria:

* Having hearing or speech impairments,
* Diagnosed with a psychotic disorder,
* Participating in another psychosocial intervention program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Increase in attitudes towards medicine in the experimental group | five week
  An increase in attitudes towards telemedicine in the experimental group compared to the pre-test measurement.

SECONDARY OUTCOMES:
no change in the control group | 5 week
  No change in the control group's attitudes towards telemedicine

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ravari, A., Sheikhoshaqi, A., Mirzaei, T., Raeisi, M., Hassanshahi, E., & Kamiab, Z. (2021). Effect of tele-nursing on blood glucose control among the elderly with diabetes: a randomized controlled trial. Evidence-Based Care, 11(2), 54-63.